CLINICAL TRIAL: NCT04049812
Title: Effectiveness of Pulse Electromagnetic Field Therapy (PEMF) on Pain, Functional Status, and Quality of Life in Patients With Chronic Radicular Pain Due to Lumbar Disc Herniation
Brief Title: Effectiveness of PEMF in Patients With Chronic Radicular Pain Due to Lomber Disc Herniation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Birkan Sonel Tur (Other)
Responsible Party: Sponsor-Investigator, Birkan Sonel Tur, Professor, Ankara University
Organization: Ankara University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 05-188-16
Record Dates: First submitted 2019-07-12; First posted 2019-08-08 (Actual); Last update posted 2019-08-08 (Actual); Status verified 2019-08

CONDITIONS: Lumbar Disc Herniation
MeSH Terms: conditions — Intervertebral Disc Displacement | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pulsed electromagnetic field (PEMF) treatment Group (Active Comparator): Group received routine hot pack, Transcutaneous electrical nerve stimulation (TENS) and PEMF treatment.
  Interventions: Device: PEMF; Device: Hot pack; Device: TENS
- Sham PEMF treatment Group (Sham Comparator): Group received routine hot pack, TENS and sham PEMF treatment.
  Interventions: Device: Hot pack; Device: TENS; Device: Sham PEMF

INTERVENTIONS:
Device: PEMF
  Arms: Pulsed electromagnetic field (PEMF) treatment Group
Device: Hot pack
Device: TENS
Device: Sham PEMF
  Arms: Sham PEMF treatment Group

SUMMARY:
The aim of this study is to investigate the effectiveness of pulse magnetic field therapy on pain, functional status, and quality of life in patients with chronic radicular pain due to lumbar disc herniation.

DETAILED DESCRIPTION:
Pulsed Electromagnetic Field Therapy (PEMF) is a non-invasive, painless treatment for various injuries, bone related conditions and pains. However, further studies on PEMF effects on low back and radicular pain is needed due to lack of studies in this area.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65
* Unilateral radicular pain for at least 3 months
* Severity of radicular pain with Visual Analog Score of at least 4/10
* Written informed consent

Exclusion Criteria:

* Pregnancy or lactation
* Cardiac pacemaker, or any metal implants or electronic devices anywhere in the body
* History of surgery or algological procedure of the lumbar region
* Physical therapy within the last year due to back pain
* Previous PEMF treatment
* Malignancy or suspicion
* Polyneuropathy (diabetic or other)
* Connective tissue disease
* Presence of inflammatory joint pain
* Fibromyalgia
* Presence of open surface wound
* Tuberculosis, mycosis, or viral disease
* Presence of pain in another region of the body with higher severity than radicular back pain
* Use of drugs other than paracetamol-derivative simple analgesics (Nonsteroidal Aanti inflammatuar, central effective, or narcotic analgesics), or less than three weeks since the discontinuation of these drugs
* Advanced mood disorder
* Radiographic evidence of Grade 2 spondylolisthesis, presence of spinal instability, and advanced degenerative spondylarthrosis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2018-03-31 (Actual)

PRIMARY OUTCOMES:
10 cm Pain Visual Analogue Scale (VAS) | 3 weeks
  The patient is asked to indicate their perceived pain intensity along a 10cm horizontal line, where '0' represents 'no pain' and '10', 'unbearable pain'.
10 cm Pain Visual Analogue Scale (VAS) | one month after treatment
  The patient is asked to indicate their perceived pain intensity along a 10 cm horizontal line, where '0' represents 'no pain' and '10', 'unbearable pain'.

SECONDARY OUTCOMES:
Disability; Roland-Morris Disability Questionnaire (RMDQ) | 3 weeks
  RMDQ has 24 yes/no questions. Scoring is between 0-24. A score of 0: no disability, score of >1 indicates disability.
Disability; Roland-Morris Disability Questionnaire (RMDQ) | One month after treatment
  RMDQ has 24 yes/no questions. Scoring is between 0-24. A score of 0: no disability, score of >1 indicates disability.
Nottingham Health Profile (NHP) | 3 weeks
  Nottingham Health Profile (NHP) is a questionnaire designed to measure a patient's view of their own health status, in a number of areas.
  The NHP consists of two parts. The first part focuses on health and comprises 38 items which deal with pain, energy, sleep, mobility, emotional reaction and social isolation. All questions have only yes/no answer options and each section score is weighted. The higher the score, the greater the number and severity of problems. The highest score in any section is 100.
Nottingham Health Profile (NHP) | One month after treatment
  Nottingham Health Profile (NHP) is a questionnaire designed to measure a patient's view of their own health status, in a number of areas.
  The NHP consists of two parts. The first part focuses on health and comprises 38 items which deal with pain, energy, sleep, mobility, emotional reaction and social isolation.All questions have only yes/no answer options and each section score is weighted. The higher the score, the greater the number and severity of problems. The highest score in any section is 100.